CLINICAL TRIAL: NCT00394368
Title: DOUBLE BLIND, MULTINATIONAL, MULTICENTRE, PARALLEL-GROUP DESIGN CLINICAL TRIAL OF THE EFFICACY AND TOLERABILITY OF CHF 1535 (BECLOMETHASONE DIPROPIONATE 100 µg + FORMOTEROL 6 µg) pMDI VIA HFA-134a vs. FLUTICASONE 125 µg + SALMETEROL 25 µg pMDI (SERETIDE®) IN THE 12-WEEK TREATMENT OF ADULT PATIENTS WITH MODERATE TO SEVERE PERSISTENT ASTHMA
Brief Title: EFFICACY AND TOLERABILITY OF BECLOMETHASONE DIPROPIONATE 100 µg + FORMOTEROL 6 µg pMDI VIA HFA-134a vs. FLUTICASONE 125 µg + SALMETEROL 25 µg pMDI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MC/PR/033011/001/03
Record Dates: First submitted 2006-10-30; First posted 2006-11-01 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Bronchial Asthma
Keywords: asthma; combinations; inhaled therapy; corticosteroids; long acting bronchodilators; salmeterol; beclomethasone; formoterol; fluticasone
MeSH Terms: conditions — Asthma | interventions — Beclomethasone; Fluticasone

INTERVENTIONS:
Drug: beclomethasone dipropionate plus formoterol fumarate combination
Drug: fluticasone propionate plus salmeterol xinafoate combination

SUMMARY:
The aim of this study was to compare the efficacy and tolerability of the fixed combination beclomethasone/formoterol pMDI with that of fluticasone/salmeterol pMDI in patients with moderate to severe asthma

DETAILED DESCRIPTION:
Asthma is a chronic disease that is estimated to affect over 25 million people both in the U.S. and Europe (i.e. approximately 10% of the total population). Pharmacological therapy is used to treat reversible airway obstruction, inflammation and hyper-reactivity. Medications include preventive treatments in forms of antinflammatory/antiallergic agents (i.e. glucocorticosteroids, leukotriene antagonists, cromolyn sodium) and reliever treatments, in form of bronchodilators (i.e. β-adrenergic agonists, anticholinergics). In patients treated with inhaled glucocorticosteroids whose asthma is not fully controlled, national and international guidelines recommend a stepwise approach. Recent evidence-based clinical trials show that the addition of a LABA to inhaled glucocorticosteroids is more beneficial in terms of asthma control than increasing the dose of corticosteroids alone.

Comparisons: CHF 1535 (BECLOMETHASONE DIPROPIONATE 100 µg + FORMOTEROL 6 µg) pMDI VIA HFA-134a compared to FLUTICASONE 125 µg + SALMETEROL 25 µg pMDI (SERETIDE®)

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of moderate to severe persistent asthma for at least 6 months, according to GINA revised version 2002 guidelines (11):

  * Forced expiratory volume (FEV1) or peak expiratory flow rate (PEFR) ³ 50% and £ 80% of the predicted normal;
  * Asthma not adequately controlled with the current therapies, defined as presence of daily asthma symptoms > once a week and night-time asthma symptoms > twice a month, and daily use of short-acting β2-agonists. These findings are to be based on recent medical history and are to be confirmed in the 2-week run-in period.
* Treatment with inhaled corticosteroids at a daily dose ≤ 1000 μg of BDP or equivalent. The daily dose of inhaled corticosteroids taken at visit 1 will be assessed taking into account the following ratios between the doses of the different steroids: fluticasone propionate : BDP CFC = 1 : 2; budesonide : BDP CFC = 4 : 5; flunisolide : BDP CFC = 1 : 1. The ratios between inhaled steroids are irrespective of the formulations (i.e. spray aerosol or powder) used. When BDP is given in the new extra-fine HFA-134a formulation (as QVAR®, 3M Healthcare), the ratio with BDP CFC is set as 2 : 5. Therefore, the maximum allowed daily dose of inhaled corticosteroids at study entry will be: budesonide 800 μg, fluticasone propionate 500 μg, flunisolide 1000 μg, BDP 1000 mg, BDP HFA extra-fine 400 μg.
* Positive response to the reversibility test in the screening visit, defined as an increase of at least 12% (or, alternatively, of 200mL) from baseline value in the measurement of FEV1 30 minutes following 2 puffs (2 ´ 100 µg) of inhaled salbutamol administered via pMDI. The reversibility test can be avoided in patients having a documented positive response in the previous 6 months.
* A co-operative attitude and ability to be trained to correctly use the metered dose inhalers and to complete the diary cards.
* Written informed consent obtained.
* At the end of the 2-week run-in period, the presence of daily asthma symptoms (of at least mild intensity) and nighttime asthma symptom (of at least mild intensity) > once a week, as well as of daily use of relief salbutamol is to be confirmed by reviewing the diary cards for run-in.

Exclusion Criteria:

* Inability to carry out pulmonary function testing;
* Diagnosis of Chronic Obstructive Pulmonary Disease (COPD) as defined by the National Heart Lung and Blood Institute/World Health Organisation (NHLBI/WHO) Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines (30);
* History of near fatal asthma;
* Evidence of severe asthma exacerbation or symptomatic infection of the airways in the previous 8 weeks;
* Three or more courses of oral corticosteroids or hospitalisation due to asthma during the previous 6 months;
* Patients treated with long-acting β2-agonists, anticholinergics and antihistamines during the previous 2 weeks, with topical or intranasal corticosteroids and leukotriene antagonists during the previous 4 weeks;
* Patients who have changed their dose of inhaled corticosteroids during the previous 4 weeks, or treatment with inhaled corticosteroids at a daily dose > 1000 μg of BDP or equivalent (except for extra-fine formulations, see inclusion criteria);
* Current smokers or recent (less than one year) ex-smokers, defined as smoking at least 10 cigarettes/day;
* History or current evidence of heart failure, coronary artery disease, myocardial infarction, severe hypertension, cardiac arrhythmias;
* Diabetes mellitus;
* Percutaneous transluminal coronary angioplasty (PTCA) or coronary artery by-pass graft (CABG) during the previous six months;
* Patients with an abnormal QTc interval value in the ECG test, defined as > 450 msec in males or > 470 msec in females;
* Other haemodynamic relevant rhythm disturbances (including atrial flutter or atrial fibrillation with ventricular response, bradycardia (≤ 55 bpm), evidence of atrial-ventricular (AV) block on ECG of more than 1st degree;
* Clinically significant or unstable concurrent diseases: uncontrolled hyperthyroidism, significant hepatic impairment, poorly controlled pulmonary (tuberculosis, active mycotic infection of the lung), gastrointestinal (e.g. active peptic ulcer), neurological or haematological autoimmune diseases;
* Cancer or any chronic diseases with prognosis < 2 years;
* Pregnant or lactating females or females at risk of pregnancy, i.e. those not demonstrating adequate contraception (i.e. barrier methods, intrauterine devices, hormonal treatment or sterilization). A pregnancy test is to be carried out in women of a fertile age.
* History of alcohol or drug abuse;
* Patients treated with monoamine oxidase inhibitors, tricyclic antidepressants or beta-blockers as regular use;
* Allergy, sensitivity or intolerance to study drugs and/or study drug formulation ingredients;
* Patients unlikely to comply with the protocol or unable to understand the nature, scope and possible consequences of the study;
* Patients who received any investigational new drug within the last 12 weeks;
* Patients who have been previously enrolled in this study;
* At the end of the run-in period, patients will not be admitted to the treatment period in the case of an increase of PEFR (L/sec) measured at the clinics at the end of the run-in period ³ 15% in respect of values measured at the start of the run-in period;
* Patients with asthma exacerbations during the run-in period will also be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 2004-11; Study Completion 2005-09

PRIMARY OUTCOMES:
morning peak expiratory flow (PEF) daily measured by patients

SECONDARY OUTCOMES:
evening PEF measured by patients daily
FEV1 measured by patients daily
standard pulmonary function tests measured at clinics at 2, 4, 8 and 12 weeks
change in FEV1 and PEF from pre-dose to 5, 15, 30 and 60 minutes after study drug intake at week 0 and 12
symptoms scores measured by patients daily
symptoms' free days measured by patients daily
use of relief salbutamol measured by patients daily
frequency of asthma exacerbations evaluated at 2, 4, 8 and 12 weeks
adverse events and adverse drug reactions daily
ECG (with QTc interval) at 0 and 12 weeks
vital signs (heart rate and blood pressure)at 2, 4, 8 and 12 weeks
12-hour (overnight)urinary cortisol/creatinine ratio at week 0 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo M. Fabbri, MD, Study Chair — Department of Respiartory Diseases - University of Modena and Reggio Emilia, Modena, Italy; Maurizio A. Vignola, MD, Study Chair — Institute of Lung Pathophysiology, National Research Council, Palermo, Italy
Locations (12):
- Poland (6):
  - Nzoz "Non nocere", Gdansk
  - Outpatients Department of Allergology "Medcare", Gdansk
  - Nzoz "Krakow Poludnie" Pulmonologic Policlinic, Krakow
  - Specialist Allergy Center All-Med, Krakow
  - Private Institute of Health and Beauty, Warsaw
  - Dolnoslaski Centre of Medical Diagnostic "Dolmed", Wroclaw
- Ukraine (6):
  - Kharkiv City Clinical Hospital 13 Pulmonological Department, Kharkiv
  - Institute of Phthisiology and Pulmonology, Academy of Medical Science of Ukraine, Depatment of Diagnostic, Therapy and Clinical Pharmacology of Lung Disease, Kiev
  - Republican Clinical Hospital Institute of Phthisiology and Pulmonology Academy of Medical Science of Ukraine, Clinical Functional Department, Kiev
  - Republican Clinical Hospital, Institute of Phthisiology and Pulmonology, Academy of Medical Science of Ukraine, Pulmonology Department, Kiev
  - Department of Hospital Therapy of Lugansk, State Medical Institute Lugansk, Regional Clinical Hospital, Luhansk
  - Department Therapy of Bronchopulmonary Pathology in Adults, Crimean Republic Research Institute of Physical Methods of Therapy and Medical Climatology, Yalta

REFERENCES:
- [Background] Gerzeli S, Rognoni C, Quaglini S, Cavallo MC, Cremonesi G, Papi A. Cost-effectiveness and cost-utility of beclomethasone/formoterol versus fluticasone propionate/salmeterol in patients with moderate to severe asthma. Clin Drug Investig. 2012 Apr 1;32(4):253-65. doi: 10.2165/11598940-000000000-00000. PMID 22352412
- [Result] Papi A, Paggiaro P, Nicolini G, Vignola AM, Fabbri LM; ICAT SE study group. Beclomethasone/formoterol vs fluticasone/salmeterol inhaled combination in moderate to severe asthma. Allergy. 2007 Oct;62(10):1182-8. doi: 10.1111/j.1398-9995.2007.01493.x. PMID 17845589
- [Derived] Oba Y, Anwer S, Maduke T, Patel T, Dias S. Effectiveness and tolerability of dual and triple combination inhaler therapies compared with each other and varying doses of inhaled corticosteroids in adolescents and adults with asthma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD013799. doi: 10.1002/14651858.CD013799.pub2. PMID 36472162